CLINICAL TRIAL: NCT05729581
Title: Effectiveness of a Reinforcement Intervention in the Breastfeeding Practice From Nutritional, Environmental and Postpartum Problem-solving Aspects to Increase the Prevalence of Breastfeeding at 6 Months Postpartum: The GREEN MOTHER Project
Brief Title: Effectiveness of Educational Intervention on Sustainable Breastfeeding: The GREEN MOTHER Project
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Parc Taulí Hospital Universitari (Other); Fundació Institut Germans Trias i Pujol (Other); Hospital de Granollers (Other); University of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 22/101-P
Record Dates: First submitted 2023-01-27; First posted 2023-02-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-03

CONDITIONS: Healthy Diet; Health Behaviour; Environmental-Pollution-Related Condition; Mothers; Child, Only
Keywords: lactation type; breastfeeding; sustainable diet; environmental impact; carbon footprint; one health
MeSH Terms: conditions — Breast Feeding | interventions — Diet, Healthy; Lactation

STUDY DESIGN:
Intervention Model Description: Our study has 2 phases: 1) observational and 2) interventional (with educational programme):
  1. st group - CG (control group) - mothers without intervention
  2. nd group - EG (experimental group) - mothers with applied educational intervention on sustainable diet and breastfeeding
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): This group of pregnant women (24-32 SG) will not be provided educational programme and information on sustainlably and healthy diet and sustainable breastfeeding. It is a control group.
- Experimental group (Experimental): This group of pregnant women (24-32 SG) will be provided educational programme and information on sustainlably and healthy diet and sustainable breastfeeding
  Interventions: Behavioral: The educational programme on sustainable and healthy diet and breastfeeding

INTERVENTIONS:
Behavioral: The educational programme on sustainable and healthy diet and breastfeeding — In the interventional group the educational programme of sustainable diet and breastfeeding will be provided before the delivery to see the impact on the prevalence of the breastfeeding at 1 and 6 months after delivery (compared with the group of control, without intervention)
  Other Names: The role of diet, products consumption, type of cooking, energy used and breastfeeding vs. artifitial lactancy in the carbon footprint
  Arms: Experimental group

SUMMARY:
Breastfeeding is the healthiest form of nutrition for the baby and is recommended to use exclusive breastfeeding (EB) until 6 months. The environmental footprint of artificial lactation (AL) has been studied, but that of EB is unknown.

Objectives:

The main objective of the first phase of the study is to identify the environmental impact in terms of the carbon footprint of breastfeeding and artificial breastfeeding, taking into account the accessories necessary for breastfeeding and of the diet and the factors associated with the diet of postpartum women in first month of life of the babies.

The main objective of the second phase is to evaluate the impact of a standardized intervention of educational programme on sustainable breastfeeding, diet and environment protection, providing inputs obtained from the first phase on the carbon footprint in the first month of life of the child and the prevalence of breastfeeding at the first month of the baby's life.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women over 16 years of age, between 24 and 32 weeks of gestation

Exclusion Criteria:

* women with a language barrier, under 16 years of age and those who do not want to participate or who do not give birth in the study associated centers

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-04-11 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Rates (number of participants, %) that use breastfeeding (exclusive) up to 6 months after the delivery | months 30-36 of the project life
  The rate of breastfeeding (exclusive) will be observed up to 6 months after the participant's baby delivery and calucalted as a percentage or fraction compared to all participants: at month of the delivery (0 month) and 1, 3 and 6 months after the delivery (giving a birth)
Rates (number of participants, %) that use EB (excusive breastfeeding) in EG (experimental group) vs. CG (group of control) | months 30-36 of the project life
  Rates (number of participants, fractions or percentages) of breasfeeding will be calculated and compared in both groups: CG (control) vs. EG (experimental).

SECONDARY OUTCOMES:
To calculate the CO2 footprint and water consumption of different types of mother diet and lactation (breastfeeding and artificial one) based on data obtained from the questionnaires | fase I) months 15-17 of the project life & phase 2) 30-36 of the project life
  Calculation (with help of the external experts) of the environmental impacts on CO2 emissions (Climate change) and water consumption (Water scarcity), using the ISO 14040 and 14044, and other related ISOs impacts of a mother's daily diet and type of breastfeeding based on data obtained from questionnaires
Assess the nutritional quality of the diet of postpartum mothers at the month of their children's life based on data obtained from the questionnaires | months 22-31 of the project life
  Assess the nutritional quality of the diet of postpartum mothers at the month of their newborn child's life: calculation of proportions of macro i micronutrients and comparison with standard recommendations (to see if the sustainable diet and breastfeeding is within healty standards or any supplementary of elements are required for it)
Comparison of rates on breastfeeding vs. artificial lactation in the population of the Northern Metropolitan area: current study results (2022/2023 based on data obtained from the questionnaire) vs. 2017 (already published) | months 30-36 of the project life
  Compare the results obtained for the rates on breastfeeding in the population of the Northern Metropolitana in the current study (2022/2023) with those obtained in 2017 (reported in the Lactem study) to see if any trends on dynamical changes in lactancy patterns are observed with time.

CONTACTS AND LOCATIONS:
Locations (1):
- ASSIR Metropolitana Nord, Sabadell, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cabedo-Ferreiro RM, Liutsko L, Cos-Busquets J, Garcia-Sierra R, Colldeforns-Vidal M, Reyes-Lacalle A, Toran-Monserrat P, Vicente-Hernandez MM, Gomez-Masvidal M, Violan C, Montero-Pons L, Falguera-Puig G, Cazorla-Ortiz G. Effectiveness of an Educational and Counseling Program (the Green Mother Project Phase 2) to Enhance Breastfeeding and Improve Mothers' Diets From an Environmental Perspective: Protocol for a Cluster Randomized Controlled Trial. JMIR Res Protoc. 2026 Jan 26;15:e80358. doi: 10.2196/80358. PMID 41587088
- [Derived] Cos-Busquets J, Cabedo-Ferreiro RM, Liutsko L, Reyes-Lacalle A, Garcia-Sierra R, Colldeforns-Vidal M, Andrade EP, Vicente-Hernandez MM, Gomez-Masvidal M, Montero-Pons L, Toran-Monserrat P, Falguera-Puig G, Cazorla-Ortiz G; GREEN MOTHER Group. A Comprehensive Assessment of the Environmental Impact of Different Infant Feeding Types: The Observational Study GREEN MOTHER. J Adv Nurs. 2025 Dec;81(12):8230-8241. doi: 10.1111/jan.16473. Epub 2024 Oct 3. PMID 39362795
- [Derived] Cabedo-Ferreiro RM, Liutsko L, Cos-Busquets J, Garcia-Sierra R, Colldeforns-Vidal M, Reyes-Lacalle A, Vicente-Hernandez MM, Gomez-Masvidal M, Montero-Pons L, Cazorla-Ortiz G, Toran-Monserrat P, Violan C, Falguera-Puig G; GREEN MOTHER Group. Environmental impact of infant feeding type, accessories used and maternal dietary habits: The GREEN MOTHER-I project, a cross-sectional study protocol. Nutr J. 2024 Aug 21;23(1):97. doi: 10.1186/s12937-024-01000-9. PMID 39164727